CLINICAL TRIAL: NCT01442415
Title: Vikings Fitness Playbook: A Family Based Lifestyle Modification Program for Overweight and Obese Youth
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to achieve enrollment goal.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1104M98872
Record Dates: First submitted 2011-08-30; First posted 2011-09-28 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle Modification (Other): Weekly 2 hour study sessions for 10 weeks; each session includes one hour of physical activity and one hour of dietary counseling
  Interventions: Behavioral: Lifestyle modification

INTERVENTIONS:
Behavioral: Lifestyle modification — Weekly lifestyle modification sessions including dietary counseling and physical activity

SUMMARY:
Childhood cancer survivors (CCS) are prone to develop obesity and are at increased risk of developing cardiovascular disease and type 2 diabetes compared to the general pediatric population. Few lifestyle modification trials have been conducted in overweight/obese CCS and it is unclear whether CCS respond similarly to lifestyle modification compared to overweight/obese individuals who have not had cancer (non-CCS). We propose a 3-year pilot study that will enroll separate cohorts of overweight/obese CCS and overweight/obese non-CCS every September into a family-based lifestyle modification program consisting of weekly sessions at the University of Minnesota. The goal of the program will be to facilitate improved physical fitness, weight management, heart health, and quality of life.

DETAILED DESCRIPTION:
Advances in cancer detection and treatment over the last few decades have led to a marked increase in survival rates in children and adolescents diagnosed with cancer. As a result, the number of CCS has burgeoned and continues to grow. Unfortunately, damage to multiple physiological systems often occurs when many of these effective, yet toxic, cancer therapies are used. In particular, radiation and chemotherapy are thought to promote an environment favorable to obesity, atherosclerosis, and impaired glucose metabolism. More specifically, the cardiometabolic risk factor profile in CCS is characterized by abdominal obesity, dyslipidemia, hypertension, and impaired glucose metabolism/insulin resistance. Excess adiposity in adolescence and young adulthood, even in otherwise healthy individuals who have not had cancer, is associated with increased risk for CVD and T2DM. Moreover, longitudinal data uniformly implicate obesity early in life as a strong predictor of future risk factor clustering and vascular abnormalities in later adulthood. Therefore, obesity in adolescence and young adulthood, even in those without a history of cancer, is associated with greatly increased risk of CVD and T2DM. The risk is likely further compounded when obesity is present in the context of cancer survivorship.

Lifestyle modification is the preferred approach for reducing the risk of developing CVD and T2DM in CCS. However, few studies have been conducted in this area and none have assessed multiple physiological outcomes. Furthermore no studies have evaluated the response to lifestyle modification in overweight/obese CCS vs. overweight/obese non-CCS. It is possible that because the cancer therapies are responsible for the increased risk in CCS (and not necessarily behavioral habits), CCS may respond less-favorably to lifestyle modification compared to overweight/obese non-CCS. Therefore, the purpose of this pilot study will be to evaluate the effect of a 10-week family-based lifestyle modification program on cardiovascular and metabolic health in overweight and obese children who have survived childhood cancers of all types and overweight and obese children who have not had cancer.

SPECIFIC AIMS

The following specific aims will be addressed in this pilot study:

1. Evaluate the effect of a 10-week family-based lifestyle modification program on physical fitness in overweight/obese children who have survived childhood cancer and overweight/obese children who have not had cancer.

   We hypothesize that compared to overweight/obese non-CCS children, overweight/obese CCS who engage in a 10-week family-based lifestyle modification program will have an attenuated improvement in peak V02.
2. Evaluate the effect of a 10-week family-based lifestyle modification program on body weight, waist circumference, blood pressure, lipids, artery health, and quality of life in overweight/obese children who have survived childhood cancer and overweight/obese children who have not had cancer.

We hypothesize that compared to overweight/obese non-CCS children, overweight/obese CCS who engage in a 10-week family-based lifestyle modification program will have attenuated improvements in body weight, waist circumference, blood pressure, lipids, artery health, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Survivor of childhood cancer for ≥5 years (N = 24) and no history of childhood cancer (N = 24)
* Age 8-16 years old at the time of consent
* BMI ≥ 85th percentile or waist circumference ≥ 85th percentile for age and gender

Exclusion Criteria:

* Exercise/physical activity contraindicated
* Initiation of a new drug therapy within the past 30 days prior to study commencement
* Current (within 3 months of study commencement) use of weight loss medication(s)
* History of weight loss surgery
* Obesity from a genetic cause (e.g., Prader-Willi)
* Central nervous system injury or severe neurological impairment
* Known systolic or diastolic dysfunction or heart failure

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change in Peak VO2 at 10 Weeks | 10 week
  Change in level of physical fitness

SECONDARY OUTCOMES:
Change in BMI at 10 Weeks | 10 week
  Change in body mass index
Change in Systolic Blood Pressure at 10 Weeks | 10 week
Change in Waist Circumference at 10 Weeks | 10 week

CONTACTS AND LOCATIONS:
Overall Officials: Aaron S. Kelly, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States